CLINICAL TRIAL: NCT01119768
Title: A Multicenter, Randomized, Open-label Phase IV Study Exploring Symptom Control Rate in Co-diagnosed NERD and Chronic Gastritis Patients Treated With 8 Weeks Esomeprazole Treatment Regimen and 2 Weeks Esomeprazole Treatment Regimen
Brief Title: Esomeprazole Treatment Co-diagnosed Non Erosive Reflux Disease (NERD) and Chronic Gastritis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9612L00127
Record Dates: First submitted 2010-04-27; First posted 2010-05-10 (Estimated); Results first posted 2012-09-28 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Non Erosive Reflux Disease; Chronic Gastritis
Keywords: GI; Nexium; Phase IV; Co-diagnosed NERD
MeSH Terms: conditions — Non-Erosive Reflux Disease | interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Esomeprazole 8 weeks treatment (Active Comparator): 20 mg q.d. (quaque die) once a day dosing for 8 weeks
  Interventions: Drug: Esomeprazole
- Esomeprazole 2 Weeks Treatment (Active Comparator): 20 mg q.d. (quaque die) once a day dosing for 2 weeks
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole — 20mg Esomeprazole once daily, 8 weeks and 24 weeks on-demand treatment
  Arms: Esomeprazole 8 weeks treatment
Drug: Esomeprazole — 20mg Esomeprazole once daily, 2 weeks and 24 weeks follow up
  Arms: Esomeprazole 2 Weeks Treatment

SUMMARY:
To compare the symptom control rate between 8 weeks esomeprazole treatment regimen group and 2 weeks esomeprazole treatment regimen group in co-diagnosed NERD and chronic gastritis patients, as evaluated by GerdQ after 24 weeks maintenance treatment/follow up.

DETAILED DESCRIPTION:
A multicenter, randomized, open-label Phase IV study exploring symptom control rate in co-diagnosed NERD and chronic gastritis patients treated with 8 weeks esomeprazole treatment regimen and 2 weeks esomeprazole treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Heartburn and/or regurgitation symptoms last for at least 3 months
* Endoscopic diagnosed as chronic gastritis (non-atrophic, and mild atrophic gastritis) within 2 weeks prior to randomization GerdQ score =8

Exclusion Criteria:

* Endoscopic visible reflux esophagitis, esophageal varices, Barrett's esophagus, malignancy or peptic ulcer Patients with Hp positive result and are eager to take Hp eradication therapy will be excluded
* If Hp positive, patients could take Hp eradication therapy after the study completion Previous PPI or H2RA therapy in the last 2 weeks before enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wenyu Guo, Study Director — AstraZeneca China MC; Prof. Yuan Yaozong, Principal Investigator — Shanghai Jiaotong University, School of Medicine, Affiliated of Ruijin Hospital
Locations (8):
- China (8):
  - Research Site, Guangzhou, Guangdong
  - Research Site, Wuhan, Hubei
  - Research Site, Nanjing, Jiangsu
  - Research Site, Jinan, Shandong
  - Research Site, Xian, Shanxi
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Beijin
  - Research Site, Shanghai

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three hundred and five patients, out of the 311 patients who signed the informed consent, were randomized to receive 8 weeks (n=154) or 2 weeks (n=151) of esomeprazole treatment.
Period: Treatment Period
Arm/Group | Esomeprazole 8 Weeks Treatment | Esomeprazole 2 Weeks Treatment
Started | 154 | 151
Completed | 136 | 126
Not Completed | 18 | 25
Not completed — Lack of Efficacy | 18 | 25
Period: Follow-up
Arm/Group | Esomeprazole 8 Weeks Treatment | Esomeprazole 2 Weeks Treatment
Started | 136 | 124
Completed | 135 | 122
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole 8 Weeks Treatment | Esomeprazole 2 Weeks Treatment | Total
Number analyzed (Participants) | 154 | 151 | 305
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 143 | 140 | 283
  >=65 years | 11 | 11 | 22
Age Continuous [Mean (Standard Deviation); unit: years] | 45.9 (12.72) | 44.9 (13.12) | 45.4 (12.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 54 | 134
  Male | 74 | 97 | 171
Region of Enrollment [Number; unit: participants]
  China | 154 | 151 | 305

OUTCOME MEASURES:

1. Primary Outcome: Symptom Control Rate at 24 Weeks Assessed by Gerd Q Questionnaire.
Description: GerdQ Scores ranging from 0 to 3 were applied for the positive predictors and from 3 to 0 (reversed order, where 3 = none) for negative predictors. The GerdQ score was calculated as the sum of these scores, giving a total score ranging from 0 to 18. When GerdQ ≥8, the patients could be symptom based diagnosed as GERD. GerdQ was consisted of 3 categories: A, B and C. Each category has two questions with sum of score ranging from 0 to 6. Symptom controlled was defined as patients with all items ≤1 in A and C category of GerdQ.
Time Frame: 24 weeks
Population: MITT was defined as patients in ITT population with symptom relief after 8 weeks or 2 weeks esomeprazole treatment
Measure: Number; unit: percentage of participants
Arm/Group | Esomeprazole 8 Weeks Treatment | Esomeprazole 2 Weeks Treatment
Number analyzed (Participants) | 136 | 126
percentage of participants | 94.9 | 87.3

2. Secondary Outcome: The Success Rate in Whole Study Duration.
Description: Success is defined as patients with symptom relief after 8 weeks or 2 weeks esomeprazole treatment, and also get symptom controlled during maintenance treatment / follow-up period.
Time Frame: 24 weeks after end of treatment
Population: Intension to Treat (ITT) was defined as all randomized subjects who took at least one dose of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Esomeprazole 8 Weeks Treatment | Esomeprazole 2 Weeks Treatment
Number analyzed (Participants) | 154 | 151
percentage of participants | 83.8 | 72.8

3. Secondary Outcome: Time to First Relapse.
Description: Time to first relapse is from the last dose during the treatment period to date of first time patient comes to the investigator due to symptom recure and need for treatment.
  Time to first relapse is actually the time when 50% of patients had relapse. Up to the end of study, there were less than 50% of the patients in arm esomeprazole 2 weeks group had relapse so was unable to compute this endpoint
Time Frame: From baseline to 24 weeks after end of treatment
Population: MITT was defined as patients in ITT population with symptom relief after 8 weeks or 2 weeks esomeprazole treatment.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Esomeprazole 8 Weeks Treatment | Esomeprazole 2 Weeks Treatment
Number analyzed (Participants) | 136 | 126
days | NA [35 to NA] — More than half of patients remained relapse free. | 57 [12 to 174]

4. Secondary Outcome: Symptom Relief Rate in 2 Treatment Regimens.
Description: Symptom relief is defined as no more than 1 day of mild symptoms of GERD during previous 7 days after 8 weeks or 2 weeks of treatment.
Time Frame: 8 weeks for arm 1, 2 weeks for arm 2
Population: ITT was defined as all randomized subjects who took at least one dose of treatment.
Measure: Number; unit: percentage of participans
Arm/Group | Esomeprazole 8 Weeks Treatment | Esomeprazole 2 Weeks Treatment
Number analyzed (Participants) | 154 | 151
percentage of participans | 88.3 | 83.4

5. Secondary Outcome: Symptom Relief Rate After 2 Weeks and 8 Weeks in 8 Weeks Treatment Group.
Description: as for outcome 4
Time Frame: 2 and 8 weeks
Population: ITT in 8 weeks treatment group
Measure: Number; unit: percentage of participants
Arm/Group | Esomeprazole 8 Weeks Treatment | Esomeprazole 2 Weeks Treatment
Number analyzed (Participants) | 154 | 0
percentage of participants
  2 weeks | 54.5 |
  8 weeks | 88.3 |

6. Secondary Outcome: Number of Patients With Unscheduled Hospital Visit(s)
Time Frame: from baseline to week 24 after end of treatment
Population: MITT
Measure: Number; unit: participants
Arm/Group | Esomeprazole 8 Weeks Treatment | Esomeprazole 2 Weeks Treatment
Number analyzed (Participants) | 136 | 126
participants | 59 | 80

7. Secondary Outcome: Percentage of Patients Satisfaction
Description: Satisfied - satisfaction score of 1-4 while very satisfied - satisfaction score of 1-2.
Time Frame: 24 weeks after end of treatment
Population: MITT
Measure: Number; unit: percentage of participants
Arm/Group | Esomeprazole 8 Weeks Treatment | Esomeprazole 2 Weeks Treatment
Number analyzed (Participants) | 136 | 126
percentage of participants
  Satisfied | 100 | 96
  Very satisfied | 48.5 | 24.6

8. Secondary Outcome: Symptom Control Rate at 8 Weeks Assessed by Gerd Q Questionnaire
Description: as for outcome 1
Time Frame: 8 weeks
Population: Modified Intension To Treat defined as patients in ITT population with symptom relief after 8 weeks or 2 weeks esomeprazole treatment
Measure: Number; unit: percentage of participants
Arm/Group | Esomeprazole 8 Weeks Treatment | Esomeprazole 2 Weeks Treatment
Number analyzed (Participants) | 136 | 126
percentage of participants | 80.1 | 75.4

9. Secondary Outcome: Symptom Control Rate at 16 Weeks Assessed by Gerd Q Questionnaire
Description: as for outcome 1
Time Frame: 16 weeks
Population: MITT was defined as patients in ITT population with symptom relief after 8 weeks or 2 weeks esomeprazole treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Esomeprazole 8 Weeks Treatment | Esomeprazole 2 Weeks Treatment
Number analyzed (Participants) | 136 | 126
percentage of participants | 85.3 | 80.2

ADVERSE EVENTS:
Time Frame: From baseline to 24 weeks after treatment.
Arm/Group | Esomeprazole 8 Weeks Treatment | Esomeprazole 2 Weeks Treatment
Serious Adverse Events (participants affected / at risk) | 0/154 | 0/151
Other Adverse Events (participants affected / at risk) | 0/154 | 0/151

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other